CLINICAL TRIAL: NCT07354932
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of SHR-2173 Injection in Patients With Primary IgA Nephropathy
Brief Title: A Study of SHR-2173 in Participants With Primary IgA Nephropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2173-205
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A: SHR-2173 injection (Experimental)
  Interventions: Drug: SHR-2173 injection
- Treatment group B: SHR-2173 injection (Experimental)
  Interventions: Drug: SHR-2173 injection
- Treatment group C: SHR-2173 injection (Experimental)
  Interventions: Drug: SHR-2173 injection
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-2173 injection — SHR-2173 injection；High dose
  Arms: Treatment group A: SHR-2173 injection
Drug: SHR-2173 injection — SHR-2173 injection；Medium dose
  Arms: Treatment group B: SHR-2173 injection
Drug: SHR-2173 injection — SHR-2173 injection；Low dose
  Arms: Treatment group C: SHR-2173 injection
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled Phase II clinical trial to evaluate the efficacy and safety of SHR-2173 in patients with Primary IgA Nephropathy(IgAN). The study consists of a screening period, a run-in period, a 48-week double-blind treatment period, and a 12-week follow-up period. Approximately 84 IgAN patients will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18 or older
2. Body weight ≥35 kg, BMI<37.5 kg/m2
3. At screening, 24-hour urinary protein quantification ≥1 g/ day, or 24-hour UPCR≥0.7 g/g
4. eGFR≥30 mL/ minute /1.73 m2 at screening
5. Female subjects with fertility or male participants whose partners are women of childbearing age must avoid donating sperm/eggs from the date of signing the ICF until 12 weeks after the last study medication, and agree to take contraceptive measures as specified in the protocol

Exclusion Criteria:

-

1、Presence of any of the following medical histories or comorbidities:

1. Renal pathology consistent with IgAN, but secondary factors could not be excluded by investigator evaluation, including but not limited to: secondary to systemic diseases, infections, autoimmune diseases or tumors;
2. A history of organ transplantation;
3. A history of splenectomy;
4. Presence or history of malignancy within 5 years before screening (note: skin squamous cell carcinoma, basal cell carcinoma or cervical carcinoma in situ with complete resection and no evidence of recurrence are excluded);
5. A history of anaphylaxis such as generalized urticaria, angioedema, or anaphylaxis, or a known history of allergy to the study drug or any component of the study drug

2、Use of any of the following drugs/treatments or participation in a clinical study:

1. Received systemic glucocorticoid therapy (including gut-targeted budesonide, etc.) within 12 weeks before randomization (Note: except those not used within 4 weeks before randomization and received prednisone ≤0.5mg/kg or equivalent glucocorticoid for non-IgAN disease within 52 weeks before randomization, with no more than 3 courses (each course ≤2 weeks);
2. Receivied immunosuppressive therapy within 12 weeks before randomization;
3. Received any investigational drug within 4 weeks before randomization or within the 5 half-lives of the trial drug, whichever was longer;
4. Received a live / attenuated live vaccine administered within 4 weeks before randomization

3、History and examination related to infection:

1. A history of infection (viral, bacterial, fungal, parasitic infection) within 3 months prior to screening, resulting in hospitalization and/or parenteral systemic antimicrobial therapy; Or a history of infection requiring systemic antimicrobial therapy within 14 days before randomization;
2. Tuberculosis (TB) or occult TB infection (one of the following conditions) :

   1. Presence of active TB or clinical symptoms of active TB at screening;
   2. Signs of active TB on imaging examination within 3 months before screening

      4、 General situation:

1) Pregnant or lactating women; 2) Investigators determine that there are circumstances that affect the safety and efficacy evaluation of the investigational drug, or other circumstances not appropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24-hour Urine Protein-to-Creatinine Ratio (UPCR) at Week 24. | Week 24.

SECONDARY OUTCOMES:
Change from baseline in 24-hour UPCR ; | up to Week 48
Change from baseline in 24-hour Urinary Albumin-to-Creatinine Ratio (UACR) ; | up to Week 48
Proportion of participants with 24-hour urinary protein quantification <0.5 g/d and <0.3 g/d ; | up to Week 48
Proportion of participants with >30% and >50% reduction from baseline in 24-hour UPCR ; | up to Week 48
Change from baseline in 24-hour urinary protein quantification ; | up to Week 48
Change from baseline in estimated Glomerular Filtration Rate (eGFR) ; | up to Week 48
Change from baseline in hematuria ; | up to Week 48
Change from baseline in serum creatinine ; | up to Week 48
Proportion of participants achieving clinical remission; | up to Week 48
Annualized total eGFR slope from baseline ; | up to Week 48
Proportion of participants meeting composite endpoints ; | up to Week 48
Change from baseline in Kidney Disease Quality of Life Short Form (KDQoL-36) ; | up to Week 48

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided